CLINICAL TRIAL: NCT05872750
Title: Rolling Deep With Gambling Disorder: From Building up of Scales, Biomarkers to Therapeutic Innovation
Brief Title: Theta Burst Stimulation for Gambling Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TCHIRB-11104005
Record Dates: First submitted 2023-05-03; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Gambling Disorder
Keywords: theta burst stimulation; Gambling Disorder
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Intervention Model Description: theta burst stimulation
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active arm (Experimental): The intervention group will receive repetitive transcranial magnetic stimulation at the left dorsolateral prefrontal cortex and pre-supplementary motor area
  Interventions: Device: theta burst stimulation
- Sham arm (Sham Comparator): the control group will receive sham stimulation
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: theta burst stimulation — Magstim Rapid 2 Plus stimulator (Magstim Co., Ltd., Whitland, United Kingdom)
  Arms: Active arm
Device: sham stimulation — sham stimulation
  Arms: Sham arm

SUMMARY:
The goal of this clinical trial is to investigate the efficacy of theta burst stimulation in individuals with gambling disorder. The main goal is to compare the severity of gambling problems following 2 weeks of intervention between active group and sham group. Participants will be randomized into active and sham group. The severity of gambling problems are assessed by self-reported questionaires.

DETAILED DESCRIPTION:
Gambling disorder, formerly known as pathological gambling, is a gambling behavior that causes significant function impairment in personal, social, occupational domains. Currently there is no pharmacological treatment for gambling disorder and it is urgent to develop innovative treatment modalities. Image studies have found a link between prefrontal circuit dysfunction and behavioral disinhibition, which supports the use of non-invasive brain stimulation as a potential treatment for gambling disorder. In this study, 75 patients with gambling disorder will be randomly assigned in a 2:1 ratio to the intervention group (50 patients) and the control group (25 patients) on double-blind basis. The study duration is 2 weeks, with 10 sessions of 20 minutes each. The intervention group will receive repetitive transcranial magnetic stimulation at the left dorsolateral prefrontal cortex and pre-supplementary motor area, while the control group will receive sham stimulation. The Chinese version of the Problem Gambling Severity Index (PGSI), the Gambling Symptom Assessment Scale (G-SAS), and the Visual Analogue Scale (VAS) for craving will be administered at week 0, 2, 4, 8, and the change in gambling severity between the two groups will be compared by repeated measures ANOVA.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 65 years;
2. fulfilling at least 4 of the Diagnostic and Statistical Manual version 5 (DSM-5) criteria of gambling disorder for at least 12-month assessed by the Structured Clinical Interview

Exclusion Criteria:

1. Inability to provide informed consent or comprehend the study procedure;
2. A major psychiatric illness that required chronic psychotropic medication or inpatient treatment, including schizophrenia spectrum disorder, bipolar spectrum disorder, and major depressive disorder with psychotic features.
3. A current DSM-5 diagnosis of substance use disorder except nicotine use disorder or the use of one to two low-potency benzodiazepine tablets for sleep impairment;
4. Have known preexisting noise-induced hearing loss, concurrent treatment with ototoxic medications, or with cochlear implants.
5. Unstable medical illness, including malignancy, uncontrolled diabetes mellitus, unstable cardiac disease or recent myocardial infarction, or cerebrovascular or cardiovascular risk factors that require intensive medical management
6. On medications known to lower seizure threshold (e.g., TCA, bupropion, clozapine)
7. Implants controlled by physiological signals, including pacemaker, implantable cardioverter defibrillator, cochlear implant.
8. Metallic objects in the head, including stenting, suture.
9. Elevated risk of seizure due to traumatic brain history, seizure history, and head trauma, intracranial lesion, and alcohol or benzodiazepines withdrawal syndrome, stimulant intoxication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in gambling craving | Before intervention (week 0) and after intervention (week 2, 4)
  Measured by visual analog scale, from 0-10
Change in gambling severity | Before intervention (week 0) and after intervention (week 2, 4)
  Measured by Gambling Symptom Assessment Scale, from 0-48

SECONDARY OUTCOMES:
Change in depression severity | Before intervention (week 0) and after intervention (week 2, 4)
  Measured by Beck Depression Inventory, from 0-63
Change in anxiety severity | Before intervention (week 0) and after intervention (week 2, 4)
  Measured by Beck Anxiety Inventory, from 0-63

CONTACTS AND LOCATIONS:
Overall Officials: Hu-Ming Chang, Principal Investigator — Taipei City Psychiatric Center, Taipei City Hospital, Taipei, Taiwan
Locations (1):
- Taipei City Hospital, Taipei, Taipei CITY, Taiwan

IPD SHARING:
Plan to Share IPD: No